CLINICAL TRIAL: NCT03150628
Title: Cytoreductive Surgery and Intraperitoneal Chemotherapy for Stomach CAncer: a Feasibility Study
Acronym: CISCA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Conflicting recruitment with PERISCOPE II study (NCT03348150)
Sponsor: Richard van Hillegersberg (Other)
Responsible Party: Sponsor-Investigator, Richard van Hillegersberg, Professor, UMC Utrecht
Organization: UMC Utrecht (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL58258.041.16; 2016-002595-27 (EudraCT Number); 16-180/G-M (Other: Ethical Review Board Number)
Record Dates: First submitted 2017-04-04; First posted 2017-05-12 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Gastric Cancer; Peritoneal Carcinomatosis; HIPEC
MeSH Terms: conditions — Stomach Neoplasms; Peritoneal Neoplasms | interventions — Cytoreduction Surgical Procedures; Hyperthermic Intraperitoneal Chemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study population (Experimental)
  Interventions: Drug: Perioperative chemotherapy; Procedure: Cytoreduction; Drug: HIPEC

INTERVENTIONS:
Drug: Perioperative chemotherapy — Perioperative chemotherapy
Procedure: Cytoreduction — Cytoreductive surgery
Drug: HIPEC — Hyperthermic intraperitoneal chemotherapy (HIPEC) with 100mg/m2 cisplatin

SUMMARY:
Rationale: For patients with peritoneal metastases of gastric origin, there is no consensus on the optimal treatment strategy. Several Asian and Western studies demonstrated hyperthermic intraperitoneal chemotherapy (HIPEC) and cytoreductive surgery (CS) to result in a prolonged survival compared to palliative systemic treatment. Morbidity and mortality rates of HIPEC and CS appear to be acceptable. In the Netherlands, this treatment is not yet introduced, therefore patients with peritoneal metastases of gastric origin are precluded from surgery and will be treated with palliative chemotherapy or best support of care.

Objective: To assess the safety and feasibility of HIPEC and CS in Western patients with peritoneal metastases of gastric cancer, in terms of morbidity and mortality. Secondary objective is to determine the effect on survival and recurrence.

Study design: Mono centre prospective phase II single-arm feasibility study.

Study population: Western patients diagnosed with resectable (cT1-4b, N1-3) gastric cancer with clinical or pathologically proven peritoneal metastases without distant metastases.

Intervention: Hyperthermic Intraperitoneal Chemotherapy (HIPEC) and Cytoreductive Surgery (CS) with Cisplatin.

Main study parameters/endpoints: Primary outcome is the safety and feasibility of the intervention, measured by the percentage of overall surgical complications grade ≥3 as stated by the Common Terminology Criteria for Adverse Events. Secondary outcomes are intraoperative events, postoperative morbidity and mortality, postoperative recovery, including quality of life, and disease free- and overall survival.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The additional burden for the patient mainly consists of HIPEC and CS.Furthermore, patients will undergo additional staging in order to exclude unresectable disease, and neoadjuvant chemotherapy regimen (3 drugs) instead of a palliative chemotherapy regimen (2 drugs). Postoperative care and outpatient visits are performed according to current protocols on HIPEC and CS for colon cancer and nation-wide protocols on gastric cancer surgery. The study is associated with a high risk classification. As there is a potential survival benefit, a small chance for curation and possibly a higher quality of life, we consider the additional burden and risks justified. This study is designed as a one group study, which eliminates group relatedness.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven adenocarcinoma of the stomach.
* Surgical resectable carcinoma (T1-4b, N1-3) (table 1)
* Pathological proven peritoneal metastases
* Peritoneal Cancer Index (PCI) ≤12
* WHO performance status 0,1 or 2 and ASA 1-3
* Age ≥ 18
* Written informed consent

Exclusion Criteria:

* Distant metastases other than peritoneal metastases
* Siewert type I/II gastro-esophageal junction tumor 22.
* Peritoneal carcinomatosis as a presentation of recurrent disease
* Pregnancy
* Any contraindication to cisplatin, e.g.

  * Hypersensitivity
  * HIV infection
  * inadequate bone marrow function (ANC <1.5x109/L or Platelets <100x109/L)
  * inadequate hepatic function (>1.5 x ULN, ALAT and ASAT >2.5 x ULN)
  * inadequate renal function (Creatinine clearance <50 ml/min)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-04-23 (Actual); Study Completion 2018-04-23 (Actual)

PRIMARY OUTCOMES:
Morbidity | From the day of surgery to hospital discharge or 30 days postoperative, whichever is last
  Common Terminology Criteria for Adverse Events (CTCAE) ≥ grade 3
Mortality | From the day of surgery to 30 days postoperative
  Postoperative mortality

SECONDARY OUTCOMES:
Survival | Up to 5 years postoperative
  Overall and disease free survival
Recovery | From the day of surgery to hospital discharge or 30 days postoperative, whichever is last
  ICU stay, hospital stay
Quality of Life | Up to 5 years postoperative
  EORTC-QLQ-C30 and EORTC-QLQ-STO22
Readmissions | Up to 30 days after hospital discharge
  Readmissions after hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Richard van Hillegersberg, MD PhD, Principal Investigator — UMC Utrecht Cancer Center, Dep. of Surgery; Jelle P Ruurda, MD PhD, Principal Investigator — UMC Utrecht Cancer Center, Dep. of Surgery
Locations (1):
- University Medical Center Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Coccolini F, Cotte E, Glehen O, Lotti M, Poiasina E, Catena F, Yonemura Y, Ansaloni L. Intraperitoneal chemotherapy in advanced gastric cancer. Meta-analysis of randomized trials. Eur J Surg Oncol. 2014 Jan;40(1):12-26. doi: 10.1016/j.ejso.2013.10.019. Epub 2013 Nov 5. PMID 24290371
- [Background] Chia CS, You B, Decullier E, Vaudoyer D, Lorimier G, Abboud K, Bereder JM, Arvieux C, Boschetti G, Glehen O; BIG RENAPE Group. Patients with Peritoneal Carcinomatosis from Gastric Cancer Treated with Cytoreductive Surgery and Hyperthermic Intraperitoneal Chemotherapy: Is Cure a Possibility? Ann Surg Oncol. 2016 Jun;23(6):1971-9. doi: 10.1245/s10434-015-5081-3. Epub 2016 Jan 11. PMID 26753751
- [Background] Glehen O, Gilly FN, Arvieux C, Cotte E, Boutitie F, Mansvelt B, Bereder JM, Lorimier G, Quenet F, Elias D; Association Francaise de Chirurgie. Peritoneal carcinomatosis from gastric cancer: a multi-institutional study of 159 patients treated by cytoreductive surgery combined with perioperative intraperitoneal chemotherapy. Ann Surg Oncol. 2010 Sep;17(9):2370-7. doi: 10.1245/s10434-010-1039-7. Epub 2010 Mar 25. PMID 20336386